CLINICAL TRIAL: NCT06646640
Title: Long Term Follow-Up Study for Individuals With Hemoglobin Disorders After Hematopoietic Cell Transplant or Gene Therapy
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEMLTFU
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hemoglobin Disorder
Keywords: Transplant; Gene Therapy
MeSH Terms: conditions — Hemoglobinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal, non-therapeutic study which includes routine assessment for long-term effects, as per FDA guidelines after receipt of an allogeneic HCT or autologous genetically modified cellular products for hemoglobin disorders.

Primary objective:

- To provide long term follow up, for individuals with hemoglobin disorders undergoing allogeneic hematopoietic stem cell transplantation (HCT) or receipt of an autologous genetically modified cellular product to treat their hemoglobinopathy. For individuals receiving a genetically modified cellular product, this long term follow up study is in accordance with the guidelines provided by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
This protocol will provide a mechanism to appropriately monitor individuals with hemoglobin disorders that have received an allogenic HCT or an autologous genetically modified cellular product for hemoglobinopathies. Monitoring will include potential long-term adverse effects after receipt of these treatments, as well as long-term monitoring after the receipt of the genetically modified cellular product.

ELIGIBILITY:
Inclusion Criteria:

* Receipt, or planned receipt, of an allogeneic HSCT or infusion of genetically modified autologous cells for hemoglobin disorders within 15 years prior to enrollment

Exclusion Criteria:

* Inability or unwillingness of research participant and/or legal guardian/ representative to provide written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 patients with hemoglobin disorders that have received, or are planning to receive, either a genetically modified cell product or allogenic HCT will be invited to enroll on this long term follow up study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
To provide ongoing review of long-term clinical and psychosocial outcomes and late effects of hematopoietic stem cell transplant and gene therapy recipients at St. Jude Children's Research Hospital. | long term follow up. Can also be stated as "up to 15 years after transplant"

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sharma, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols